CLINICAL TRIAL: NCT02580760
Title: Circulating Silicone After Cosmetic Silicone Injection in Transgender Patients
Brief Title: Transgender, Silicone and Blood Smear
Acronym: TSBS
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: 15FBT-TSBS
Record Dates: First submitted 2015-09-30; First posted 2015-10-20 (Estimated); Last update posted 2016-01-25 (Estimated); Status verified 2015-09

CONDITIONS: Injection; Complications, Sepsis; Injection Site Disorder; Injection Site Extravasation; Intentional Poisoning by Silicone
Keywords: Silicone; Transgender; Dermatology; Blood contamination; Adverse event after injection
MeSH Terms: conditions — Sepsis; Injection Site Reaction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cosmetic silicone injection: People responding to inclusion criteria with a history of cosmetic silicone injection

SUMMARY:
This cross-sectional monocentric study will describe transgender men transitioning into women and who had cosmetic silicone injection.

The principal objective is to estimate the prevalence of Transgender with circulating monocytes containing silicone vacuoles in blood smears among Male to Female Transgender population with a history of cosmetic silicon injections.

The secondary objectives are to describe the transgender population, to describe the quantity of silicone in vacuoles of circulating monocytes, and the association between dermatological complications (inflammatory and not inflammatory) and several clinical and biological characteristics (HIV status, level of immunosuppression, inflammatory syndrome, quantity of silicone which was injected , silicone quantity in blood smears).

DETAILED DESCRIPTION:
Injectable liquid silicone is a permanent filling product which is no more used in France because of a high risk of complications. Cosmetic silicone injection is a common feminization approach for transgender populations.

This cross-sectional monocentric study will describe transgender men transitioning into women and who had cosmetic silicone injection.

The principal objective is to estimate the prevalence of Transgender with circulating monocytes containing silicone vacuoles in blood smears among Male to Female Transgender population with a history of cosmetic silicon injections.

The secondary objectives are to describe the transgender population, to describe the quantity of silicone in vacuoles of circulating monocytes, and the association between dermatological complications (inflammatory and not inflammatory) and several clinical and biological characteristics (HIV status, level of immunosuppression, inflammatory syndrome, quantity of silicone which was injected , silicone quantity in blood smears).

ELIGIBILITY:
Inclusion Criteria:

* Adults
* Not in opposition to data collection
* Transgender men transitioning into women patients with cosmetic silicone injection
* Consultation in Bichat hospital

Exclusion Criteria:

* Unable to communicate
* Guardianship, curatorship

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Every transgender men transitioning into women patients with cosmetic silicone injection and consulting in Bichat hospital.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2015-07; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
The prevalence of Transgender with circulating monocytes containing silicone vacuoles in blood smear among Male to Female Transgender population, the day of their consultation. | 1 day ,the day of their consultation
  The prevalence of Transgender with circulating monocytes containing silicone vacuoles will be calculated as the number of subjects with monocytes containing silicone vacuoles in blood smears on the number of subjects with a history of silicone cosmetic injection

SECONDARY OUTCOMES:
Number of monocytes with vacuoles of silicone in a standardized area of 25 monocytes per blood smear slide | 1 day ,the day of their consultation
Size of silicone vacuoles in monocytes | 1 day ,the day of their consultation
Inflammatory and not inflammatory dermatological complications | 1 day ,the day of their consultation
  assessment of dermatological complications during the clinical examination
Number of patients with a positive HIV status | 1 day ,the day of their consultation
  Number of patients with a positive HIV status
Level of immunosuppression estimated with viral charge | 1 day ,the day of their consultation
  HIV viral load, the day of the admission or the last value known in the 6 month prior to the consultation
Level of immunosuppression estimated with cluster of differentiation 4 cell (CD4) rate | 1 day ,the day of their consultation
  CD4 cell count the day of the consultation or the last value known in the 6 month prior to the consultation.
  CD4 cell stands for Cluster of differentiation antigen 4 cell.
Inflammatory syndrome estimated with C-reactive protein (CRP) | 1 day ,the day of their consultation
Inflammatory syndrome estimated with ferritin | 1 day ,the day of their consultation
Amount of injected silicone, in liters | 1 day ,the day of their consultation
Time since the first silicone injection for cosmetic purposes, in years | 1 day ,the day of their consultation
Comorbidities: Number of patients with history of Tuberculosis | 1 day ,the day of their consultation
  Number of patients with history of Tuberculosis
Comorbidities: Number of patients with history of Hepatitis B | 1 day ,the day of their consultation
  Number of patients with history of Hepatitis B
Comorbidities: Number of patients with history of Hepatitis C | 1 day ,the day of their consultation
  Number of patients with history of Hepatitis C
Comorbidities: Number of patients with history of Syphilis | 1 day ,the day of their consultation
  Number of patients with history of Syphilis

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice Bouscarat, MD, Study Director — Hôpitaux Universitaires Paris-Nord Val de Seine, site Bichat
Locations (1):
- Hôpitaux Universitaires Paris-Nord Val de Seine, site Bichat, Paris, France